CLINICAL TRIAL: NCT06611527
Title: Comparison Between Two Methods of Positive Pressure Therapy in the Prevention of Pulmonary Complications in the Immediate Postoperative Period of Cardiac Surgery: a Prospective, Randomized Clinical Trial
Brief Title: Positive Pressure Therapy to Optimize LUNG Function After Heart Surgery
Acronym: PRO-LUNGHS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Marcia Souza Volpe, Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RPPI
Record Dates: First submitted 2024-09-18; First posted 2024-09-25 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Period; Physical Therapy Modalities; Continuous Positive Airway Pressure; Respiratory Function Tests; Pulmonary Atelectasis; Heart Surgery
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PS+PEEP group (Active Comparator): PS+PEEP modality involves the application of two levels of positive pressure intermittently.
  Interventions: Device: PS+PEEP group
- CPAP group (Experimental): Continuous positive airway pressure modality.
  Interventions: Device: CPAP group

INTERVENTIONS:
Device: PS+PEEP group — Application of 4 sets of 20 repetitions with PS to provide a tidal volume equal to 10ml/kg of predicted body weight, PEEP equal to 10 cmH2O, and inspired oxygen fraction (FiO2) to achieve peripheral oxygen saturation (SpO2) between 92-94%
  Arms: PS+PEEP group
Device: CPAP group — Application of CPAP of 10 cmH2O with FiO2 to achieve SpO2 between 92-94% for 30 minutes.
  Arms: CPAP group

SUMMARY:
The most common cardiac surgeries are myocardial revascularization and valve replacement or plastic surgery. In the postoperative period of cardiac surgeries, the incidence of pulmonary complications ranges from 30% to 50% and is associated with increased length of hospital stay and morbidity and mortality. To reduce or minimize the occurrence of these complications, respiratory physiotherapy employs positive pressure reexpansion therapies, such as continuous positive airway pressure (CPAP) and positive pressure support with positive end-expiratory pressure (PS+PEEP).

The goal of this clinical trial is to compare the effects of two positive pressure therapies, CPAP versus PS+PEEP, on the incidence of pulmonary complications in patients in the postoperative period of myocardial revascularization and valve replacement or plastic surgery, with mild to moderate pulmonary dysfunction.

The main question it aims to answer is: Do patients in the immediate postoperative period of myocardial revascularization or valve replacement/plastic surgery, exhibiting mild to moderate pulmonary dysfunction, experience a comparable reversal of pulmonary conditions when treated with PS+PEEP versus CPAP?

Participants will undergo the following assessments: spirometry, respiratory muscle strength testing, handgrip strength testing, and electrical impedance tomography.

In the immediate postoperative period, participants will be randomized into two treatment groups: • Control Group PS+PEEP - application of 4 sets of 20 repetitions with PS to provide a tidal volume equal to 10ml/kg of predicted body weight, PEEP equal to 10 cmH2O, and inspired oxygen fraction (FiO2) to achieve peripheral oxygen saturation (SpO2) between 92-94%; • Experimental Group CPAP - application of CPAP at 10 cmH2O with FiO2 to achieve SpO2 between 92-94% for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Immediate postoperative period of myocardial revascularization and/or valve replacement or plastic surgery;
* Patients in the preoperative period at risk of developing pulmonary complications, characterized by the presence of at least 2 of the following risk factors: age ≥ 70 years, productive cough, diabetes, history of smoking, chronic obstructive pulmonary disease (COPD) defined by forced expiratory volume in 1 second (FEV1) lower than 75% of predicted, body mass index (BMI) ≥ 27 kg/m2, or only FEV1 lower than 80% and FEV1/forced vital capacity (FVC) ratio lower than 70% of predicted; OR patients in the postoperative period (up to 12 hours after extubation) with mild to moderate complications characterized by a pulmonary complication score lower than 3.

Exclusion Criteria:

* Hemodynamic instability characterized by mean arterial pressure (MAP) lower than 60mmHg and/or acute arrhythmia of any etiology;
* Need for intra-aortic balloon;
* Duration of invasive mechanical ventilation exceeding 24 hours after surgery;
* Pulmonary complication score ≥ grade 3;
* Presence of signs of acute respiratory failure, such as respiratory rate (f) ≥ 25 breaths/min and use of accessory muscles;
* Chest tube with air leak;
* Use of a pacemaker or implantable or external cardioverter-defibrillator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Severity of pulmonary complications in the postoperative period | Participants will be followed for 7 days after surgery.
  Score of pulmonary complications adapted from previous publications, with 5 degrees, where the higher one (5) means death before hospital discharge, and degree 4 means need of invasive mechanical ventilation due to acute respiratory failure.
Electrical impedance tomography (EIT) ventilation distribution | EIT ventilation distribution will be monitored during and 30 minutes after the therapies.

SECONDARY OUTCOMES:
Length of ICU stay | From the day of surgery up to ICU discharge, an expected average of 2 days, and maximum censoring at day 28 after surgery.
Length of hospital stay | From the day of surgery up to hospital discharge, an expected average of 10 days, and maximum censoring at day 28 after surgery.
Handgrip strength | Assessments will be conducted preoperatively, on the 5th and 7th postoperative days.
Maximal inspiratory and expiratory pressures | Assessments will be conducted preoperatively, on the 5th and 7th postoperative days.
Spirometry test results | Spirometry will be conducted preoperatively, on the 5th and 7th postoperative days.
  Forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), and the FEV1/FVC ratio from the spirometry test will be presented as percentages of predicted values.
Positive pressure therapy comfort level | The level of comfort will be evaluated immediately after the first three positive pressure therapy sessions.
  Comfort during positive pressure therapy will be assessed using a visual analog scale ranging from 0 to 10, where 0 represents maximum comfort and 10 represents extreme discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia S Volpe, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Instituto do Coração - HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
IPD will be stored at https://domusdados.unifesp.br/ All IPD that results in a publication will be shared upon reasonable request.
Supporting Information: Study Protocol
Time Frame: IPD will be avaible from 12 months to 36 months after publication.